CLINICAL TRIAL: NCT06957158
Title: The Effect of Serum Calcium Levels on Postoperative Pain in Patients Undergoing Abdominal Surgery: A Prospective Observational Study
Brief Title: The Effect of Serum Calcium Levels on Postoperative Pain: A Prospective Observational Study
Status: Recruiting | Type: Observational
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Serum calcium levels and pain
Record Dates: First submitted 2025-04-26; First posted 2025-05-04 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-04

CONDITIONS: Postoperative Pain
Keywords: Serum calcium levels; Postoperative pain; Ionized calcium levels
MeSH Terms: conditions — Pain, Postoperative | interventions — Arterial Pressure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood and arterial blood were collected
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Peripheral venous blood — Peripheral venous blood was collected before and after the surgery to measure the total serum calcium levels.
Diagnostic Test: Arterial blood — Arterial blood was collected before anesthesia induction and after removal of the artificial airway to measure ionized calcium levels.

SUMMARY:
This is a prospective observational study. To investigate the effect of serum calcium levels on postoperative pain in patients undergoing abdominal surgery, and to determine whether changes in serum calcium levels are a risk factor for postoperative pain.

DETAILED DESCRIPTION:
This study aimed to measure the total serum calcium and ionized calcium levels both before and after surgery. Additionally, NRS scores were recorded at different time points.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years old
* American Society of Anesthesiologists Classification I-III
* Patients undergoing elective abdominal surgery under general anesthesia
* Patients participate voluntarily and sign an informed consent form

Exclusion Criteria:

* Patients with a history of severe disease
* Patients with chronic preoperative pain and/or long-term analgesic use
* Patients with hearing disorders or verbal communication difficulties
* Patients with psychiatric disorders or cognitive dysfunction
* Patients requiring mechanical ventilation or ICU admission after surgery
* Patients with a history of substance or alcohol abuse Patients who could not cooperate with the study for any reason

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent elective abdominal surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of pain NRS score ≥6 within 48 hours after surgery | From the end of the surgery to 48 hours after surgery
  NRS score: pain was assessed using a 10-point NRS (range: 0-10, 0 and 10 indicate no pain and the most extreme pain imaginable, respectively）

SECONDARY OUTCOMES:
The maximum incisional pain score at 0-12h postoperatively | From the end of the surgery to 12 hours after surgery
  NRS score: pain was assessed using a 10-point NRS (range: 0-10, 0 and 10 indicate no pain and the most extreme pain imaginable, respectively）
The maximum incisional pain score at 12-24h postoperatively | From 12hours to 24 hours after surgery
  NRS score: pain was assessed using a 10-point NRS (range: 0-10, 0 and 10 indicate no pain and the most extreme pain imaginable, respectively）
The maximum incisional pain score at 24-48h postoperatively | From 24 hours to 48 hours after surgery
  NRS score: pain was assessed using a 10-point NRS (range: 0-10, 0 and 10 indicate no pain and the most extreme pain imaginable, respectively）
The maximum visceral pain score at 0-12h postoperatively | From the end of the surgery to 12 hours after surgery
  NRS score: pain was assessed using a 10-point NRS (range: 0-10, 0 and 10 indicate no pain and the most extreme pain imaginable, respectively）
The maximum visceral pain score at 12-24h postoperatively | From 12 hours to 24 hours after surgery
  NRS score: pain was assessed using a 10-point NRS (range: 0-10, 0 and 10 indicate no pain and the most extreme pain imaginable, respectively）
The maximum visceral pain score at 24-48h postoperatively | From 24 hours to 48 hours after surgery
  NRS score: pain was assessed using a 10-point NRS (range: 0-10, 0 and 10 indicate no pain and the most extreme pain imaginable, respectively）
Whether additional analgesia was administered within 48 hours after surgery | From the end of the surgery to 48 hours after surgery
  The proportion of patients who received additional analgesia out of the total patient group
Patient-controlled intravenous analgesia opioid consumption | From the end of the surgery to 24 hours and 48 hours after surgery
  PCIA opioid consumption was assessed by checking the PCIA electronic system

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data for this study is available from the sponsor on reasonable request through email
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Five years after the study